CLINICAL TRIAL: NCT06040372
Title: Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Compound LB54640 in Healthy Overweight and Obese Subjects
Brief Title: A First in Human Study to Assess the Safety, Tolerability of LB54640 in in Healthy Overweight and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-MCCL001
Record Dates: First submitted 2023-08-21; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Obese; Overweight; Healthy
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: This was a randomized, double-blind, placebo-controlled study conducted in two parts. Study Part 1 had a SAD design to investigate the safety, tolerability, and PK of LB54640 administered orally in healthy overweight and obese subjects. Study Part 1 included a cohort (Cohort S3) to assess the effect of food on LB54640, which was conducted with a blinded, placebo-controlled, two-way crossover design. Study Part 2 had a MAD design to investigate the safety, tolerability, PK, and PD of LB54640 administered orally in healthy overweight and obese subjects
Who Masked: Participant, Investigator
Masking Description: Double blind, there will be unblinded pharmacist for investigational product distribution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LB54640 (Experimental): 5 mg, 25 mg and 200 mg strengths
  Subjects will be administered once daily and duration vary per each cohorts.
  Single Ascending Dose (SAD) cohorts : 1 day
  * SAD 1 10mg
  * SAD 2 25mg
  * SAD 3 50mg (Food effect cohort)
  * SAD 4 100mg
  * SAD 5 200mg
  * SAD 6 400mg
  healthy Multiple Ascending Dose (MAD) cohorts: 28days
  * MAD 1 10mg
  * MAD 2 25mg
  * MAD 3 50mg
  * MAD 4 100mg
  * MAD 5 200mg
  * MAD 6 400mg
  * MAD 7 600mg
  Interventions: Drug: LB64640
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB64640 — The investigational product (IP) LB54640 is provided 5 mg, 25 mg and 200 mg strengths.
  Arms: LB54640
Drug: Placebo — Placebo is provided as a matching placebo
  Arms: Placebo

SUMMARY:
The aim of this 4-weeks randomized double-blind placebo-controlled single and multiple ascending dose study is to assess the Safety and Tolerability of LB54640 in Healthy overweight and obese subjects

DETAILED DESCRIPTION:
The study was conducted in 2 parts:

Part 1 (Single Ascending Dose) This study part included 6 sequential dose cohorts (S1-S6), enrolling 8 healthy subjects per cohort. Cohort S3 was evaluate the effect of food.

Part 2 (Multiple Ascending Dose) This part included 7 sequential dose cohorts (M1-M7), enrolling 8 subjects per cohort. Cohorts was evaluate safety, Pharmacokinetics and Pharmacodynamics parameters in healthy overweight and obese subjects. They were dosed once daily for 28 days with LB54640 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 to ≤ 70 years.
* Body mass index (BMI) ≥ 27 kg/m2, with stable body weight by history for 3 months (defined as change < 5%)
* HbA1c < 6.5%.
* Female subjects must be non-pregnant and non-lactating. Females of childbearing potential must use at least two of the medically accepted contraceptive methods, table at least 4 weeks prior to the screening.
* Ability to provide written informed consent.

Exclusion Criteria:

* History or current diagnosis with T1DM or T2DM.
* History or current diagnosis of any malignancy.
* History of pheochromocytoma or insulinoma.
* History or current diagnosis of cardiac dysrhythmias or heart disease
* History of surgical treatment for obesity or any other gastrointestinal surgery
* History of major depression, anxiety, suicidal behavior or attempts, or other psychiatric disorder.
* Use of approved weight-lowering pharmacotherapy
* Has a clinically significant history of suicidal ideation or suicidal behavior as assessed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Through study completion upto 6weeks depending on cohorts
  Number of subjects who experienced adverse events and severity of adverse events
Incidence and severity of adverse events of special interest (AESIs) in Part 2 (MAD) | Through study completion upto 6weeks depending on cohorts
  Number of subjects who experienced adverse events of special interest (AESIs)
Change from baseline in vital signs (blood pressure) | Through study completion upto 6weeks depending on cohorts
  Absolute values and changes from baseline (BP assessed by 24-hour ambulatory blood pressure monitoring (ABPM);systolic pressure and diastolic pressure will be assessed
Change from baseline in vital signs (heart rate) | Through study completion upto 6weeks depending on cohorts
  Absolute values and changes from baseline (HR assessed by 24-hour ambulatory electrocardiography monitoring (12-lead cardiac telemetry; central reader))
Change from baseline in vital signs (weight in kilograms, height in meters) | Through study completion upto 6weeks depending on cohorts
  weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Pharmacokinetics profiles in Plasma for single ascending dose cohort | Through study completion upto 1week
  Peak Plasma Concentration (Cmax) during the dosing periods
Pharmacokinetics profiles in Plasma for single ascending dose cohort | Upto 1week
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetics profiles in Plasma for single ascending dose cohort | Through study completion upto 1week during the single ascending dose cohort
  Terminal half-life (t1/2)
Pharmacokinetics profiles in urine for single ascending dose cohort | upto 1week
  Renal clearance (CLR)
Pharmacokinetics profiles in urine for single ascending dose cohort | Through study completion upto 1week depending on cohorts
  Amount of unchanged drug excreted into urine (Ae) for specific collection intervals
Pharmacokinetics profiles in plasma for multiple ascending dose cohort | upto 2weeks
  Maximum concentration (Cmax)
Pharmacokinetics profiles in plasma for multiple ascending dose cohort | Through study completion upto 2weeks
  Area under the concentration-time curve (AUC) during the dosing periods

OTHER OUTCOMES:
Effect of food by Pharmacokinetics profiles | Through study completion upto 1week
  Area under the concentration-time curve (AUC) (total and various incremental AUCs, including AUClast, AUC0-infinity)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Mirza, Principal Investigator — Clinical Research Unit
Locations (1):
- Clinical Research Unit, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No